CLINICAL TRIAL: NCT03377621
Title: Whole Body Vibration for Obstructive Sleep Apnea
Brief Title: Whole Body Vibration for OSA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not funded, and therefore not conducted
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Mary A. Woo, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-001323
Record Dates: First submitted 2017-12-06; First posted 2017-12-19 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: whole body vibration; sleep; apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea

STUDY DESIGN:
Intervention Model Description: One group will receive intervention and will be evaluated before and after intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Whole Body Vibration (Experimental): OSA subjects will be asked to use whole body vibration machine for 30 minutes, 3 times a week for 6 weeks in between visits.
  Interventions: Device: Whole Body Vibration

INTERVENTIONS:
Device: Whole Body Vibration — Whole Body Vibration Machine from the company Confidence Fitness

SUMMARY:
Obstructive Sleep Apnea (OSA) is a serious medical condition which is increasing in the United States and significantly increases risks for other diseases, morbidity and mortality. The most common treatment for OSA is CPAP (Continuous Positive Airway Pressure), but this intervention has low patient compliance, significant expense ($800-2,000/set), and high inconvenience. Whole Body Vibration (WBV) training is a novel OSA intervention which could have higher patient compliance, low expense, and potentially lower morbidity and mortality and improved quality of life in this increasing patient population.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) can be defined as temporary cessation of breathing (often from 10-30 seconds) during sleep caused by a blockage of the airways. OSA is increasing in the United States and currently afflicts at least 18 to 25 million adults in the country. OSA is a chronic disease which increases the risk of hypertension, heart disease, Type 2 diabetes, stroke, and depression. OSA also has negative effects on the brain, such as significant reductions in white matter and gray matter, which are accompanied by impairments to cognition, mood, and daytime alertness. At this time, the most common and effective way to treat OSA is with the use of continuous positive airway pressure (CPAP).

Adequate CPAP usage (use of the CPAP mask/device for at least 4 hours/night for a minimum of 70% of the nights = 5 days/week) is associated with higher sleep quality, increased daytime alertness, improved mood, better memory, decreased blood pressure, greater cardiac left ventricular ejection fraction, and decreased dysrhythmias. Yet despite the significant benefits of CPAP, compliance (use of CPAP for at least 4 hours per night for at least 5 out of 7 nights/week) with CPAP continues to be low (17-54%). Terri Weaver Predictors of CPAP non-compliance are unclear, but most researchers and clinicians cite OSA patient dislike for the equipment (lots of tubing, sometimes noisy), mask discomfort, and inconvenience. Alternatives to CPAP, such as uvuloectomy and dental jaw devices, are either invasive or have less efficacy in some OSA subjects. One non-invasive method to treat OSA which has not been reported in the literature is whole body vibration (WBV).

Whole body vibration refers to any vibration of any frequency which is transferred to the human body. Theoretically, WBV creates eccentric muscle reaction and enables anaerobic activity and was initially designed as a form of resistance training. WBV has been used as a successful treatment for osteoporosis, stroke, leg muscle strength and balance in the elderly. However, it has never been utilized or suggested as a treatment for OSA. In a pilot study conducted by the investigators, they found that 30 minutes of WBV (using a commercially available device which costs $250), 3 times per week, for 6 weeks, dramatically decreased apnea-hypopnea index (AHI; a measure of sleep-disordered breathing) in persons with moderate to severe OSA without changes in weight or injury and that WBV treatment compliance was very good.

Yet why would WBV have any impact on OSA? According to the investigators' early studies, stimulation of the proprioception nerves (neural system which allows sensorimotor location of the limbs) stimulates the apneustic center of the lower pons (top of spinal cord), which in turn promotes respiratory inspiration. In the investigators' other studies, they have demonstrated that stimulation of the proprioception nerves during sleep stimulates breathing. However, one might ask if WBV is not being administered during sleep, but only while awake, why would this impact breathing during sleep? It appears that respiratory training while awake continues to have impact during sleep, as witnessed by the fact that such activities as opera singing, trumpet or didgeridoo instrument playing, have been used to successfully treat OSA. The investigators theorize that these activities (including WBV) entrain breathing and thus "condition" the apneustic center to improve airway dilation during sleep. Despite the promising preliminary data, the impact of WBV needs to be examined in a larger number of persons with OSA and the neural mechanisms of WBV on the apneustic regions of the lower pons remain to be explored.

ELIGIBILITY:
Inclusion Criteria:

* Must be between ages 21-60
* Clinical diagnosis of moderate-to-severe OSA (AHI > 15)
* Must be able to stand up for 30 mins at a time with no joint or muscular problems
* Must have adequate space/power in home to run the WBV machine

Exclusion Criteria:

* Previous history of stroke and/or myocardial infarction
* Diagnosed neuropsychological and neuropsychiatric diseases,
* Airway or chest deformities that would interfere with breathing,
* Chronic obstructive pulmonary disease,
* Cystic fibrosis
* Presence of brain mass lesions
* Any history of drug abuse (e.g., cocaine or tobacco)
* History of renal failure (requiring dialysis).
* Pregnancy (if female) due to the potential dangers to the fetus from the MRI
* Subjects with contraindications to MRI:

  * Metallic and electronic implants (phrenic or cardiac pacemakers), braces, or metallic-based tattoos
  * Body weight > 275 pound
  * Claustrophobia
* Inadequate space/ electronic power in home to run the WBV machine.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-02 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline OSA Severity at 6 weeks | Baseline and 6 weeks
  OSA severity as measured by Apnea-Hypopnea Index (AHI)
Change from Baseline Brain Structure at 6 weeks | Baseline and 6 weeks
  Brain structure as measured by brain magnetic resonance imaging

SECONDARY OUTCOMES:
Change from Baseline PSQI at 6 weeks | Baseline and 6 weeks
  Sleep quality as measured by Pittsburgh Sleep Quality Index (PSQI)
Change from Baseline Nonin Wristox Measurement at 6 Weeks | Baseline and 6 weeks
  Sleep quality as measured by Nonin Wristox2
Change in Baseline Balance at 6 weeks | Baseline and 6 weeks
  Balance as measured by timing how long subject can balance on dominant foot (in seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Woo, PhD, RN, Principal Investigator — UCLA School of Nursing
Locations (1):
- 300 Medical Plaza, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share all de-identified (i.e., no personal identifiers or other HIPAA-related information) data
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available 6 months after study completion
Access Criteria: Applicant must e-mail the principal investigator to request access and must submit specific aims and data analysis plans for the information. Applicant must have an academic e-mail (i.e., affiliated with a research academic institution, such as an accredited university or research agency - examples: NIH, RAND Corporation, University of Pennsylvania, etc)

REFERENCES:
- [Background] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Background] Castronovo V, Scifo P, Castellano A, Aloia MS, Iadanza A, Marelli S, Cappa SF, Strambi LF, Falini A. White matter integrity in obstructive sleep apnea before and after treatment. Sleep. 2014 Sep 1;37(9):1465-75. doi: 10.5665/sleep.3994. PMID 25142557
- [Background] Billings ME, Auckley D, Benca R, Foldvary-Schaefer N, Iber C, Redline S, Rosen CL, Zee P, Kapur VK. Race and residential socioeconomics as predictors of CPAP adherence. Sleep. 2011 Dec 1;34(12):1653-8. doi: 10.5665/sleep.1428. PMID 22131602
- [Background] Weaver TE, Grunstein RR. Adherence to continuous positive airway pressure therapy: the challenge to effective treatment. Proc Am Thorac Soc. 2008 Feb 15;5(2):173-8. doi: 10.1513/pats.200708-119MG. PMID 18250209
- See also: National Healthy Sleep Awareness Project — http://www.sleepeducation.org/healthysleep